CLINICAL TRIAL: NCT05592366
Title: Adapting and Testing the Care Partner Hospital Assessment Tool for Use in Dementia Care
Brief Title: Dementia Care Partner Hospital Assessment Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-0352; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 10/29/2024 (Other: UW Madison); 1K23AG080068-01 (NIH)
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Participants in this arm will only receive standard of care.
- Adjusted CHAT-AD (Experimental): Using CHAT, participants will be asked questions about their needs to fully support and care for their loved one after the loved one is released from the hospital.
  Interventions: Behavioral: Care Partner Hospital Assessment Tool

INTERVENTIONS:
Behavioral: Care Partner Hospital Assessment Tool — Complete the adjusted CHAT as well as demographic and caregiving questionnaires during and after loved one's hospitalization.
  Arms: Adjusted CHAT-AD

SUMMARY:
The purpose of this study is to see whether an adapted questionnaire called the Care Partner Hospital Assessment Tool (CHAT) for care partners of hospitalized patients living with Alzheimer's disease and related dementias (ADRD) (CHAT-AD) can help people with dementia receive better care after they go home from the hospital. Participants will be a care partner ('family member or friend') who provides unpaid care to a hospitalized adult relative or partner to help them take care of themselves because of dementia. Participants can expect to be in this study for 14 days.

DETAILED DESCRIPTION:
The purpose of this study is to adapt CHAT for care partners of hospitalized patients living with ADRD (CHAT-AD) and evaluate its feasibility and potential efficacy in a pilot randomized clinical trial. Findings from this study will enable the lead researcher to launch an independent program of research that aims to (1) improve hospital-based care processes and outcomes for patients living with ADRD and their care partners, and (2) make clear the essential caregiving role that so many care partners of patients living with ADRD assume.

In order to adapt CHAT, there will be two design teams with key stakeholders from local aging networks and a large academic medical system: one team comprised of previously hospitalized patients living with ADRD and their care partners (N=7 dyads) and the second comprised of healthcare system administrators and clinicians (N=7). The team will use a validated participatory human-centered design process in which each team completes 5 co-design videoconference sessions that occur in parallel across 4 months, with 2-3 weeks between each session.

Upon adaptation of the CHAT-AD, the study team will partner with a medical and surgical units that are part of a large academic medical system to recruit 128 eligible care partners of hospitalized patients living with ADRD, randomized into either the CHAT-AD plus usual care or usual care-only groups. The team will assess feasibility by examining overall recruitment, attrition, safety, adherence, and implementation satisfaction. To examine efficacy, a validated measure of caregiving preparedness will be obtained pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provide unpaid care to a hospitalized adult relative or partner to help them take care of themselves because of ADRD
* 18 years or older

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Preparedness for Caregiving | Baseline to 72 hours post-discharge
  Using the Preparedness for Caregiving Scale, which is a self-rated assessment that consists of eight items that asks care partners how well prepared they believe they are for multiple domains of caregiving, change in preparedness will be measured. Preparedness is defined as perceived readiness for multiple domains of the caregiving role such as providing physical care, providing emotional support, setting up in-home support services, and dealing with the stress of caregiving. Responses are rated on a 5-point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score the more prepared the care partner feels for caregiving.
Care partner satisfaction of care | 72 hours post-discharge
  The Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) is a 29-item survey that asks discharged patients about their recent hospital stay. The study team will modify and use three items from this survey to capture care partner satisfaction of care. These items are rated on a 4-point case from 1 (definitely no or strongly disagree) to 4 (definitely yes or strongly agree), with higher scores representing more care partner satisfaction with care.

SECONDARY OUTCOMES:
Feasibility measure: Time to complete assessments and CHAT-AD | Baseline
  The actual amount of time taken to complete the assessments and CHAT-AD will be recorded in study records.
Qualitative Feasibility measure: Adherence | 72 hours post-discharge
  Participants will self-report the reasons for not having followed the CHAT-AD protocol.
Change in care partner burden | Baseline to 72 hours post-discharge
  The Zarit Burden Interview is a self-rated assessment that consists of 22 items that asks care partners about their burden related to the care they provide a relative. Responses are rated on a 5-point scale with scores ranging from 0 (never) to 4 (nearly always). The Zarit Burden Interview score is obtained by adding the score for each question (total points). The higher the score the more burden the care partner feels.
Change in care partner depression | Baseline to 72 hours post-discharge
  The Patient Health Questionnaire-2 (PHQ-2) is a self-rated assessments that consists of 2 items that asks care partners about the frequency of depressed mood and anhedonia over the past two weeks. Responses are rated on a 4-point scale with scores ranging from 0 (not at all) to 3 (nearly every day). The PHQ-2 score is obtained by adding the score for each question (total points). The higher the score the more depressed the care partner feels. A score of 3 can be used as the cutpoint when screening for depression.
Feasibility measure: Implementation satisfaction | 72 hours post-discharge
  Clinician questionnaire composed of 5 Likert questions (scale of 1-5) as well as open-ended questions. A higher number on the Likert scale indicates higher satisfaction.
Post-treatment Qualitative Interviews: Attrition | 72 hours post-discharge
  Qualitative analysis will proceed concurrently with data collection to allow identified themes related to attrition to be explored in subsequent interviews. All team members will analyze the data and look for themes and trends that are emergent from the data.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Fields, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fields B, Werner N, Shah MN, Hetzel S, Golden BP, Gilmore-Bykovskyi A, Farrar Edwards D. Adapting and Testing the Care Partner Hospital Assessment Tool for Use in Dementia Care: Protocol for a 2 Sequential Phase Study. JMIR Res Protoc. 2023 Jun 22;12:e46808. doi: 10.2196/46808. PMID 37347517